CLINICAL TRIAL: NCT02472444
Title: Etude du contrôle hédonique de la Prise Alimentaire Par l'Analyse Des Potentiels évoqués Gustatifs
Brief Title: Gustatory Evoked-related Potentials in Humans
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: GEP
Record Dates: First submitted 2015-06-01; First posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Gustatory Evoked Potentials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Taste perception plays an important role in maintaining nutritional balance. Gustatory evoked potentials (GEP) can be detected in response to an intermittent stimulation of the gustatory receptors by a primary flavour. GEP are non invaisve, painless and safe.

The aims were to establish a reliable recording of GEP in Humans and to determine physiological variations of the gustatory evoked cerebral activity, by recording gustatory evoked potentials in different physiological situations (different intensities of taste solutions, after feeding or fasting, with different taste...). Healthy volunteers were included in this study. GEP were recorded in 9 cortical sites by EEG sensors (10/20 system), in front of the primary and the secondary gustatory cerebral areas, referenced against ear lobes.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* non smoker

Exclusion Criteria:

* diabetes mellitus
* treatment interfering with taste
* history or current neurological problem

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy young volunteers
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
latencies of the gustatory evoked potentials | during a 20 minutes taste stimulus
amplitudes of the gustatory evoked potentials | during a 20 minutes taste stimulus

REFERENCES:
- [Derived] Jacquin-Piques A, Gaudillat S, Mouillot T, Gigot V, Meillon S, Leloup C, Penicaud L, Brondel L. Prandial States Modify the Reactivity of the Gustatory Cortex Using Gustatory Evoked Potentials in Humans. Front Neurosci. 2016 Jan 5;9:490. doi: 10.3389/fnins.2015.00490. eCollection 2015. PMID 26778949